CLINICAL TRIAL: NCT02537938
Title: A Randomized, Placebo-Controlled, Double-blind, Parallel-Group, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Orally-administered NGP 555 in Healthy Subjects
Brief Title: Neurogenetic Pharmaceuticals (NGP) 555 in Healthy Volunteers (14 Day Multiple Ascending Dose)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroGenetic Pharmaceuticals Inc (Industry)
Collaborators: WCCT Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NGP 555-002
Record Dates: First submitted 2015-08-26; First posted 2015-09-02 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NGP 555 (Experimental): NGP 555 given once a day for 14 days as a capsule; 100 mg, 200 mg, or 400 mg
  Interventions: Drug: NGP 555
- Placebo (No Intervention): Placebo comparator given once a day for 14 days as a capsule.

INTERVENTIONS:
Drug: NGP 555
  Arms: NGP 555

SUMMARY:
This study involves the use of an investigational drug called NGP 555. In each group of healthy subjects, 2 people will receive placebo and 6 people will receive NGP 555.

DETAILED DESCRIPTION:
The purpose of this research study is to determine the safety, tolerability, and pharmacokinetics (PK) of multiple (14 days), oral doses of NGP 555 in healthy volunteers.

NGP 555 has been created for the treatment of Alzheimer's disease (AD). NGP 555 is being developed to prevent Abeta 42 amyloid formation, a protein that is likely a key factor in the development of AD.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female volunteers aged 40-65 yrs and in good health as determined by medical history, physical examination, clinical laboratory studies, electrocardiograms (ECGs), vital signs, and investigator judgement
2. Volunteer voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB)-approved informed consent prior to performing any of the screening procedures
3. Female volunteers who are post-menopausal or surgically sterile
4. Female volunteers who are of child-bearing potential must agree to use a medically acceptable method of contraception
5. Male healthy volunteers willing to use barrier contraception (i.e., condoms) even if their partners are post-menopausal, surgically sterile or are using acceptable contraceptive methods
6. Body mass index (BMI) of ≥ 18.0 kg/m2 to ≤ 32.0 kg/m2

Exclusion Criteria:

1. Personal history of seizure disorder, symptomatic seizures (not including a history of simple febrile seizures in childhood) or any past or present medical condition which, in the opinion of the investigator has the potential to reduce seizure threshold (e.g., history of head trauma or concussion, previous alcohol abuse, substance abuse)
2. Any concurrent disease or condition that, in the opinion of the Investigator, would make the volunteer unsuitable for participation in the clinical study
3. Volunteer has history of alcohol and/or illicit drug abuse within two years of entry
4. Any psychiatric diagnosis or symptoms (e.g., hallucinations, major depression, anxiety or delusions)
5. History of cerebrovascular events or non-vasovagal related loss of consciousness
6. History of cardiac arrhythmias, ischemic heart disease, cerebrovascular disease.
7. Hepatic impairment as defined by >1.3 times the upper limit of normal ranges of serum liver enzymes
8. Renal impairment as defined by >1.3 abnormal ranges of serum creatinine
9. Abnormal blood pressure
10. Abnormal cardiovascular parameters
11. Volunteers with abnormally low serum B12, folate or abnormal thyroid function tests
12. Positive Screening test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody, or human immunodeficiency virus (HIV) antibody
13. Positive urine test for alcohol or drugs
14. Any suicidal behavior in the last 2 years
15. Female volunteers that are breastfeeding or female volunteers with a positive urine pregnancy test
16. Volunteers unwilling to avoid consumption of coffee and caffeine containing beverages
17. Unable to abstain from smoking (or other nicotine use)
18. Donation of blood (> 500 mL) or blood products within 2 months
19. Volunteers who take prohibited medications
20. Use of an investigational drug within 30 days prior to Screening (Visit 1)
21. Unwilling to abstain from vigorous exercise
22. Clinically significant deviation from normal in physical examination, vital signs or clinical laboratory tests
23. Volunteer is unable to understand the protocol requirements, instructions and study-related restrictions, the nature, scope and possible consequences of the clinical study
24. Volunteer is unlikely to comply with the protocol requirements, instructions and study-related restrictions (e.g., uncooperative attitude, inability to return for follow-up visit and improbability of completing the clinical study)
25. Volunteer has medical conditions that are unstable or which, in the clinical opinion of the Investigator, may interfere with study procedures or volunteer safety. Volunteers with the following stable medical conditions, adequately controlled with stable doses of concomitant medications, need not be excluded if in the opinion of the Investigator, their conditions do not compromise volunteer safety or study procedures:

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of adverse events or safety outcomes | Baseline to 23 days
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Apinya Vutikkilaird, DO, Principal Investigator — WCCT
Locations (1):
- WCCT Global, Cypress, California, United States